CLINICAL TRIAL: NCT00132444
Title: Phase I Study of the Safety and Acceptability of UC-781 Topical Vaginal Microbicide in Heterosexual Women and Their Male Partners
Brief Title: Study of UC-781 Vaginal Microbicide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: Emory University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: CONRAD, CONRAD
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4413
Record Dates: First submitted 2005-07-11; First posted 2005-08-22 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV; topical microbicides
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): 0.25% gel
  Interventions: Drug: topical vaginal application of UC-781 gel
- 2 (Active Comparator): 0.1% gel
  Interventions: Drug: topical vaginal application of UC-781 gel
- 3 (Placebo Comparator)
  Interventions: Drug: topical vaginal application of UC-781 gel

INTERVENTIONS:
Drug: topical vaginal application of UC-781 gel — UC-781 gel (arms 1 and 2) or placebo (arm 3) applied vaginally twice daily for 14 days

SUMMARY:
This study will help determine whether the agent UC-781, formulated as a gel, is safe when applied to the vagina twice daily for 14 days. It will also assess whether women find the gel acceptable to use.

DETAILED DESCRIPTION:
Purpose: To assess the safety and acceptability of vaginal use of 0.1% and 0.25% UC-781 gel in sexually active HIV-uninfected women, and their male partners, and sexually abstinent HIV-infected women

Design: Single-center, phase I randomized, double-blind, controlled trial with 14 days of twice-daily product or control gel exposure

Study population: Sexually active, HIV-uninfected women at low-risk for HIV and their male partners; sexually-abstinent HIV-infected women; all age 18-45

Size: 36 sexually active HIV-uninfected women and up to 36 of their male partners; 18 sexually abstinent HIV-infected women

Treatment regimen:

Stage 1: HIV-uninfected, sexually active women and 1 male partner per woman:

12 women assigned to 0.1% UC-781 twice daily x 14 days; 12 women assigned to 0.25% UC-781 twice daily x 14 days; 12 women assigned to control gel twice daily X 14 days.

Stage 2: HIV-infected, abstinent women: 12 assigned to 0.25% UC-781 twice daily x 14 days; 6 assigned to control gel twice daily x 14 days

Study duration: Participant accrual will take 6 months. Each participant will be followed for 14 days in Stage 1 and 21 days in Stage 2. Total study duration will be 9 months.

Study Site: The Hope Clinic of Emory University, Decatur, GA

Primary Objectives:

* To assess the safety and toxicity of 0.1% UC-781 gel and 0.25% UC-781 gel administered intravaginally twice-daily for 14 days on the vulvar and cervicovaginal mucosa of sexually active HIV-uninfected women
* To assess the safety and toxicity of 0.25% UC-781 gel administered intravaginally twice-daily for 14 days on the vulvar and cervicovaginal mucosa of sexually abstinent HIV-infected women

Secondary Objectives:

* To assess the acceptability of 0.1% and 0.25% UC-781 gel administered intravaginally twice-daily for 14 days among HIV-uninfected, and the acceptability of 0.25% gel similarly administered to HIV-infected women
* To assess the effect of study product on vaginal microflora of HIV-uninfected and HIV-infected women
* To assess the systemic absorption of 0.1% and 0.25% UC-781 gel when administered intravaginally
* To assess HIV viral load in genital secretions in HIV-infected women during 0.25% UC-781 gel use
* To assess the genotypic resistance patterns of HIV in genital secretions and peripheral blood in HIV-infected women during 0.25% UC-781 gel use
* To assess the acceptability of 0.1% and 0.25% UC-781 gel in male sexual partners of HIV-uninfected women

Primary Endpoints:

The safety and toxicity of 0.1% UC-781 gel and 0.25% UC-781 gel administered intravaginally twice-daily for 14 days in sexually-active HIV-uninfected women and 0.25% UC-781 gel administered in sexually-abstinent HIV-infected women will be assessed by:

* Macroscopic and/or microscopic evidence of vulvar and/or vaginal epithelium damage, including ulceration, abrasion, severe erythema, and/or severe edema
* Macroscopic and/or microscopic evidence of cervical mucosal damage including ulceration, abrasion, severe erythema, and/or severe edema
* Symptoms of genital irritation, including burning, itching or soreness
* Laboratory evidence of grade 3 or higher toxicity for hematology, liver or renal function which cannot be attributed to another cause

Secondary Endpoints:

Acceptability of 0.1% and 0.25% UC-781 gel use by HIV-uninfected and 0.25% UC-781 gel use by HIV-infected women will be assessed by:

* Proportion of participants who at Day 14 visit indicate they would be 'somewhat unlikely' or 'very unlikely' to use 0.1% and 0.25% UC-781 gel during sexual intercourse in the future compared to control gel users
* Reported positive aspects of using 0.1% and 0.25% UC-781 gel compared to control gel users
* Reported negative aspects of using 0.1% and 0.25% UC-781 gel compared to control gel users

ELIGIBILITY:
Inclusion Criteria:

For All Females:

* Ages 18-45 years of age
* Able to provide written informed consent
* Normal Pap smear at screening or documentation of such within six months prior
* Regular monthly menses or amenorrhea due to hormonal contraceptive use
* Agree to pelvic exam, colposcopy and biopsy (if indicated) per protocol
* Able/willing to complete Study Diary
* Agree to abstain from sexual intercourse for 48 hours prior to the enrollment visit
* Agree to apply assigned study gel as required per protocol
* Agree to abstain from the following activities from at least 48 hours prior to enrollment through the Day 14 visit:

  * Insertion of fingers/objects into the vagina
  * Receiving oral sex
  * Receiving anal sex
  * Using a diaphragm, cervical cap, female condom, or vaginal contraceptive ring
  * Using vaginal products other than the study gels
  * Participating in other vaginal microbicide or contraceptive studies

Additional Inclusion Criteria for Stage 1:

* HIV-uninfected
* In a monogamous sexually active relationship with one male partner throughout the study
* Report having vaginal intercourse only with that partner at least two times per week
* Agree to use study-provided male condoms for each act of vaginal intercourse while taking part in the study
* Agree to inform male partner about participation

Additional Inclusion Criteria for Stage 2:

* HIV-infected
* Sexually abstinent or agree to abstain from sexual intercourse while taking part in the study
* Under regular medical care for HIV management
* CD4+ lymphocyte count > 200/mm3 for the last 6 months
* HIV viral load > 4.0 log10 copies/ml at screening
* Documentation of prior HIV genotype with one or more mutations conferring resistance to a non-nucleoside reverse transcriptase inhibitor (NNRTI)
* Not currently on antiretrovirals
* Willing to provide study staff with access to medical records related to their HIV infection

Inclusion Criteria for Male Partners:

* Ages 18 years or older
* Able to give written informed consent
* Male sexual partners of HIV-uninfected women taking part in Stage 1 of the study

Exclusion Criteria:

Exclusion Criteria for All Females:

* Are post-menopausal
* Have had a hysterectomy
* Clinically significant chronic medical condition (other than HIV) that is considered progressive.
* History of malignancy, with the exception of basal cell or squamous cell skin cancer
* Pregnant or planning to become pregnant in the next three months
* Currently breastfeeding
* History of sensitivity or allergy to latex or any compound used in this study
* Have received antibiotics in the 14 days prior to enrollment
* Have used a spermicide or spermicidally lubricated condom within 7 days prior to enrollment
* Have been using a hormonal contraceptive method for less than 3 months prior to enrollment
* Have participated in other microbicide or contraceptive studies in the past three months
* Grade 3 or higher liver, renal or hematology abnormality, as defined by the Table for Grading the Severity of Adult Adverse Events at screening
* Have a positive bacterial urine culture
* Currently have a clinically detectable genital abnormality (i.e. vulvar, vaginal, cervical and/or perineal ulcer or lesions or abnormal Pap smear)
* In the three months prior to enrollment have had any of the following:

  * An abnormal Pap smear
  * A pregnancy
  * An abortion
  * An intrauterine device (IUD)
  * Breakthrough menstrual bleeding
  * Vaginal bleeding during or following vaginal intercourse
  * Gynecologic surgery
  * Signs consistent with a sexually transmitted disease (STD)
  * Signs of genital trauma
  * Signs of genital tract infection other than asymptomatic bacterial vaginosis (BV)
* In the six months prior to enrollment have had any of the following:

  * History of treatment for or a diagnosis with a new STD
  * Exchanged sex for money, drugs or gifts
  * Protected (with condoms) penile-vaginal or penile-anal sexual contact with more than 4 partners
  * Unprotected (without condoms) penile-vaginal or penile-anal sexual contact with more than 1 partner
  * A male sexual partner who was diagnosed or treated for an STD (other than HIV)
  * A male sexual partner who has injected drugs
* Are currently using, or in the last year have used intravenous drugs (except for therapeutic use), crack or other recreational drugs
* Are currently abusing, or in the last year have abused alcohol.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Additional Exclusion Criteria for Stage 1:

* Unprotected (without condoms) or protected (with condoms) penile-vaginal or penile-anal sexual contact with an HIV-infected partner in the past 6 months
* Unwilling to use study-provided male condoms while on study

Additional Exclusion Criteria for Stage 2:

* NNRTI mutations in plasma and/or genital secretions at screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Macroscopic and/or microscopic evidence of cervical, vulvar and/or vaginal epithelial damage, including ulceration, abrasion, severe erythema, and or severe edema. | with two weeks of administration
Symptoms of genital irritation, including burning, itching or soreness | With 2 weeks of administration
Laboratory evidence of grade 3 or higher toxicity for hematology, liver or renal function which cannot be attributed to another cause | with 2 weeks of administration

SECONDARY OUTCOMES:
Acceptability of 0.1% and 0.25% UC-781 gel use by HIV-uninfected and HIV-infected women | queried after 2 weeks of administation

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Workowski, MD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic of Emory University, Decatur, Georgia, United States